CLINICAL TRIAL: NCT04900259
Title: The Effect of the COVID-19 Pandemic on Primary Bladder Cancer Presentations
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: COVIDBC2021
Record Dates: First submitted 2021-05-23; First posted 2021-05-25 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Bladder Cancer; Covid19
Keywords: Bladder cancer; COVID-19; Transurethral resection
MeSH Terms: conditions — Urinary Bladder Neoplasms; COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Bladder Cancer: Patients diagnosed with primary bladder cancer in the COVID-19 period
  Interventions: Behavioral: COVID-19 pandemic
- PreCOVID-19 Bladder Cancer: Patients diagnosed with primary bladder cancer in the preCOVID-19 period
  Interventions: Behavioral: COVID-19 pandemic

INTERVENTIONS:
Behavioral: COVID-19 pandemic — Patients diagnosed with primary bladder cancer by transurethral resection in the urology clinic during and before the COVID-19 pandemic will be retrospectively evaluated and compared.

SUMMARY:
In this study, investigators aim to reveal how the COVID-19 pandemic process affects primary bladder cancer presentations, tumor stages and degrees, the time elapsed between diagnosis and intervention, tumor recurrence and progression, which are oncological results.

DETAILED DESCRIPTION:
The rapid spread of the 2019 coronavirus disease (COVID-19) caused by a novel betacoronavirus known as the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) has had dramatic effects on individuals and health systems around the world. Beyond those infected with SARS-CoV-2, the intense demand for limited health system resources has led to reduced capacity, rapid depletion of healthcare systems, and hospitals becoming a source of virus transmission.

Urology associations and reference centers have issued recommendations to inform urology care during the COVID-19 outbreak. It is essential that urologists give priority to patient safety. Potential delays in the diagnosis and treatment of urological conditions and the additional burden on healthcare resources must be balanced against the risks of exposure to COVID-19. While this situation aims to conserve healthcare resources, it has created the risk of delaying cancer treatment. As a result, the transformation of health services and the increasing interest of the public in avoiding exposure to the disease has led to a decrease in the number of hospital admissions.

The effects of the pandemic on patients with bladder cancer due to a decrease in emergency room and urology clinic admissions are not clear. During the COVID-19 outbreak, the EAU (European Association of Urology) panel of non-muscle invasive bladder cancer published an evidence-based guideline. According to this guideline, four priority groups were formed and a certain period of delaying treatment was defined for patients in each group according to their priorities.

ELIGIBILITY:
Inclusion Criteria:

* Primary bladder cancer

Exclusion Criteria:

* Previous history of urinary tract tumor
* Chronic kidney disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with primary bladder cancer by transurethral resection in the urology clinic.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-15 (Actual)

PRIMARY OUTCOMES:
Rate of tumor stages | 2 months
  Rate of tumor stages in patients who diagnosed with bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kaan Yildiz, Principal Investigator — Ankara Training and Resarch Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heldwein FL, Loeb S, Wroclawski ML, Sridhar AN, Carneiro A, Lima FS, Teoh JY. A Systematic Review on Guidelines and Recommendations for Urology Standard of Care During the COVID-19 Pandemic. Eur Urol Focus. 2020 Sep 15;6(5):1070-1085. doi: 10.1016/j.euf.2020.05.020. Epub 2020 Jun 5. PMID 32532703
- [Background] Esperto F, Pang KH, Albisinni S, Papalia R, Scarpa RM. Bladder Cancer at the time of COVID-19 Outbreak. Int Braz J Urol. 2020 Jul;46(suppl.1):62-68. doi: 10.1590/S1677-5538.IBJU.2020.S107. PMID 32549074
- [Background] Wallis CJD, Novara G, Marandino L, Bex A, Kamat AM, Karnes RJ, Morgan TM, Mottet N, Gillessen S, Bossi A, Roupret M, Powles T, Necchi A, Catto JWF, Klaassen Z. Risks from Deferring Treatment for Genitourinary Cancers: A Collaborative Review to Aid Triage and Management During the COVID-19 Pandemic. Eur Urol. 2020 Jul;78(1):29-42. doi: 10.1016/j.eururo.2020.04.063. Epub 2020 May 3. PMID 32414626